CLINICAL TRIAL: NCT05720572
Title: Clinical Efficacy and Safety of Antazoline in Comparison to Propafenone in Conversion of Paroxysmal Atrial Fibrillation to Sinus Rhythm - a Single Center, Randomized, Double-blinded Study (the AnProAF Study).
Brief Title: Antazoline in Comparison to Propafenone in Pharmacological Cardioversion of Atrial Fibrillation.
Acronym: AnProAF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Jarosław Karwowski, Principal Investigator, Centre of Postgraduate Medical Education
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMKP/85/PB/2019
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Atrial Fibrillation
Keywords: Antazoline; Antiarrhythmic drugs; Pharmacological cardioversion; Atrial fibrillation; Randomized controlled trial
MeSH Terms: conditions — Atrial Fibrillation | interventions — Antazoline; Propafenone

STUDY DESIGN:
Intervention Model Description: Study design This randomized, double-blind, placebo-controlled, non-inferiority clinical study is actually carried out at the Department of Heart Disease, Centre of Postgraduate Medical Education, Warsaw, Poland. The study will include 390 participants presenting with an episode of AF lasting less than 48 h. All participants must sign an informed consent form.
  The study protocol was approved by the local ethics committee and is in full compliance with the Declaration of Helsinki.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: After eligible patients provide informed consent, they are assigned a specific identifier. Neither the patient nor the researcher knows which group the subject will be assigned to. Patients are randomized according to the implemented random allocation sequence using numbered sealed envelopes, which are opened after inclusion of the patient for the study in a 1:1 ratio to treatment with antazoline or propafenone.
  After inclusion of the patient the study the nurse will open the numbered envelope and prepare three 10 cm3 syringes with study drugs according to randomization and pass them to the enrolling physician and nurse who will administer the drug.
  The patient, enrolling physician, nurse who administering the drug, and clinician reviewing the clinical outcomes will all be blinded to the treatment. The statistician, study nurse who prepares the syringes and clinician involved in safety control will be unblinded to the patient's assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antazoline (Experimental): Any patient fulfilling the inclusion criteria will be prepared to pharmacological cardioversion in a standard way comprising of standard baseline 12-lead ECG, continuous ECG monitoring, periodic noninvasive blood pressure monitoring (BP) and iv line.
  After drug administration the patient will be observed for 3 hours after the first dose with exit ECG and BP measure taken at the end of observation. Further treatment of the patient depends on clinical state and follows appropriate clinical guidelines.
  Interventions: Drug: Antazoline
- Propafenone (Active Comparator): Any patient fulfilling the inclusion criteria will be prepared to pharmacological cardioversion in a standard way comprising of standard baseline 12-lead ECG, continuous ECG monitoring, periodic noninvasive blood pressure monitoring (BP) and iv line.
  After drug administration the patient will be observed for 3 hours after the first dose with exit ECG and BP measure taken at the end of observation. Further treatment of the patient depends on clinical state and follows appropriate clinical guidelines.
  Interventions: Drug: Propafenone

INTERVENTIONS:
Drug: Antazoline — Participants assigned to the antazoline group will be administered antazoline in boluses in boluses of 100 mg diluted to 20 cm3 every 10 minutes up to a total dose of 300 mg diluted to 60 cm3 or conversion of AF to SR. Drug administration will also be stopped in case of an adverse event or conversion of AF to a different supraventricular arrhythmia. BP will be measured before every injection.
  Arms: Antazoline
Drug: Propafenone — Patients assigned to the propafenone group were administered three 20-cm3 boluses every 10 minutes up to 60 cm3 or conversion of AF to SR. Each of the first two boluses included 70 mg propafenone (total dose 140 mg), and the third bolus contained only 20-cm3 0.9% NaCl. Drug administration will be stopped in case of an adverse event or conversion of AF to a different supraventricular arrhythmia. BP will be measured before every injection.
  Arms: Propafenone

SUMMARY:
The purpose of this randomized, double blind, non-inferiority clinical trial was to compare the clinical efficacy and safety of antazoline with propafenone in the rapid conversion of paroxysmal non-valvular atrial fibrillation to sinus rhythm in patients without heart failure

DETAILED DESCRIPTION:
Background

Atrial fibrillation (AF) is the most common type of arrhythmia, and occurs in approximately 3% of the population over 20 years of age and 9% of those over 80 years of age [1]. Restoration of sinus rhythm (SR) remains an integral part of the treatment for this type of arrhythmia. Early pharmacological (PCV) or electrical cardioversion (ECV) is necessary to improve symptoms, prevent the side effects of the prolonged crisis of arrhythmia, and avoid hospitalization. ECV requires general sedation and does not prevent from immediate AF recurrence. Therefore, the majority of patients are qualified for pharmacological attempts to terminate the arrhythmia. The early PCV of AF to SR may be achieved by administration of Class (Vaughan-Williams) IA, IC, and III antiarrhythmic drugs (AADs): flecainide, ibutilide, dofetilide, propafenone, amiodarone, or novel agent vernakalant. These AADs have limitations such as proarrhythmic side effects in patients with structural heart disease (IC), delayed onset of action (amiodarone), high cost, and low availability (vernakalant) [1].

An efficacious, well-tolerated, less expensive antiarrhythmic drug with rapid onset of action is necessary. Antazoline meslate is an antihistaminic agent with antiarrhythmic quinidine-like properties, which have been documented in 1960s [2,3]. Electrophysiologically, antazoline prolongs action potential duration and lowers its amplitude, prolongs phase-0 duration, reduces phase-4 of resting potential, and reduces excitability of cardiac tissue. Anticholinergic action of this drug leads to transient increase of heart rate, improving atrioventricular conduction and increasing the corrected QT-interval, left atrial refractory period, and inter-atrial conduction time [4-6]. In human healthy volunteers, the terminal elimination half-life of antazoline was 2.29 hours with a mean residence time of 3.45 hours [7]. In clinical practice, the drug can be administered intravenously in boluses of 50-100 mg every 3-5 minutes until successful cardioversion or up to a cumulative dose of 250-350 mg [8].

In Poland, it was registered for intravenous termination of supraventricular arrhythmias. Unfortunately, antazoline is not listed in any of the formal guidelines due to the lack of large randomized trials comparing this drug with other AADs in SR restoration. To the best of our knowledge, only one randomized clinical trial has been published that evaluated the antiarrhythmic effect of antazoline in comparison to placebo [9]. In antazoline group (38 patients), successful conversion of AF to SR was achieved in 72.2%, with a median duration of 16 minutes. Other published observational studies have shown high efficacy of antazoline, ranging between 50% and 80% and a rapid onset of action with cardioversion duration between 7 and 20 minutes [3,8,10-14]. The aim of this randomized, double blind, placebo-controlled, non-inferiority clinical trial is to assess clinical efficacy of antazoline in rapid conversion of atrial fibrillation to sinus rhythm in patients with paroxysmal atrial fibrillation without significant valvular disease or advanced heart failure.

Methods Study objectives The purpose of the study is to assess clinical efficacy of antazoline in rapid conversion of AF to SR in comparison to propafenone in patients with paroxysmal atrial fibrillation without significant valvular disease or advanced heart failure. Due to a presumed lack of statistical power, secondary end points and safety analysis will be considered exploratory.

Study design This randomized, double-blind, placebo-controlled, non-inferiority clinical study is actually carried out at the Department of Heart Disease, Centre of Postgraduate Medical Education, Warsaw, Poland. The study will include 390 participants presenting with an episode of AF lasting less than 48 h. All participants must sign an informed consent form. Approval for the study was obtained from the local ethics committee (nr 85/PB/2019; July 10, 2019).

The study protocol was approved by the local ethics committee and is in full compliance with the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for participating in the study and written standard version of informed consent for cardioversion accepted at the Department of Heart Disease, Warsaw, Poland
* Age 18 to 90years
* AF lasting < 48 hours
* Stable cardio-pulmonary state on enrollment
* In case of unclear history of heart failure or suspicion of left ventricle damage echocardiographyis indicated prior to enrollment

Exclusion Criteria:

* Lack of written informed consent
* Allergy to antazoline or propafenone
* Intolerance of anatzoline or propafenone
* AF related to significant valvular disease
* Clinically significant heart failure or ejection fraction <50%
* Systolic blood pressure (BP) <100 mmHg
* History of significant bradyarrhythmia not treatedwith permanent pacemaker
* Resting ventricular rate of < 80 bpm without pacemaker backup
* Heart rate > 140 bpm
* Tachycardia >160'
* Advanced liver or kidney failure
* Acute coronary syndrome, coronary artery by-passgraft, stroke or transient ischemic attack within 30 days before enrollment
* Preexcitation in ECG not treated by radiofrequency ablation of accessory pathway
* Signs and symptoms of ischemia related to AF
* An investigational drug used within 30 days before enrollment
* Advanced liver or kidney failure
* QT prolongation over 440 ms or QTc (Bazett's formula) over the population norm
* Pregnancy or breast feeding
* Background therapy of any oral AADs.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Conversion of atrial fibrillation (AF) to sinus rhythm (SR) | 3 hours
  Conversion of AF to SR confirmed in standard 12-lead ECG during the observation period

SECONDARY OUTCOMES:
Time to conversion of atrial fibrillation to sinus rhythm | 3 hours
Serious adverse event defined as every adverse event requiring hospitalization or prolonged observation | 3 hours
Disturbances of atrioventricular conduction | 3 hours
Hypotension < 90mmHg | 3 hours
Pauses > 4s | 3 hours
  Pauses in heart beat
Tachycardia > 180bpm | 3 hours
Nausea and/or vomiting | 3 hours
Hot flush | 3 hours
Drowsiness | 3 hours
Headache | 3 hours
Bitter/metallic taste | 3 hours
Anxiety | 3 hours
New complex ventricular arrhythmia | 3 hours
Prolongation of QTc in ms (Bazett's formula) in comparison to baseline | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jarosław JK Karwowski, PhD, Principal Investigator — Centre of Postgraduate Medical Education
Locations (1):
- Postgraduate Medical School, Warsaw, Poland